CLINICAL TRIAL: NCT05157386
Title: Physical Exercise as Adjunctive Therapy for Affective Disorder and Anxiety - a Retrospective Study of the Braining Project 2017-2020 Regarding Feasibility, Participants and Changes in Symptoms, Function and Physical Parameters
Brief Title: Physical Exercise as Adjunctive Therapy for Affective Disorder and Anxiety
Status: Active, not recruiting | Type: Observational
Sponsor: Region Stockholm (Other Government)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Sponsor
Other Study IDs: Braining Study 1 Retrospective
Record Dates: First submitted 2021-11-09; First posted 2021-12-15 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Depression; Physical Inactivity; Bipolar Disorder; Anxiety Disorders; Anxiety; Posttraumatic Stress Disorder; ADHD; Autism; Social Phobia; Panic Disorder; Generalized Anxiety Disorder; Personality Disorders; Insomnia; Stress
Keywords: physical exercise; training; physical activity; treatment
MeSH Terms: conditions — Depression; Sedentary Behavior; Bipolar Disorder; Anxiety Disorders; Stress Disorders, Post-Traumatic; Attention Deficit Disorder with Hyperactivity; Autistic Disorder; Phobia, Social; Panic Disorder; Generalized Anxiety Disorder; Personality Disorders; Sleep Initiation and Maintenance Disorders; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants in Braining, years 2017-2020: Braining was primarily open for patients with a main or secondary diagnosis within affective disorder or anxiety syndromes, sleep disturbance or stress.
  Participants in Braining (n≈600), who have participated in three or more training sessions 2017-2020 (n≈250), and who agree to contribute to this study, will be included.
  Interventions: Other: Braining

INTERVENTIONS:
Other: Braining — Core components of Braining: Personnel-led training sessions, motivating contact with psychiatric staff, measurement and evaluation before and after the training period; usually 12 weeks. PE is added on to treatment as usual (TAU). The training sessions are moderate to intense aerobic group training, 30-45 minutes. Each training session is preceded by a short (5-10 minutes) individual meeting with staff including assessment of daily form, motivational work, and the opportunity to ask questions. The target frequency for participation is preferably at least three training sessions/week during a 12 week period. The training period for each patient begins with an informative and motivating group or individual lecture or and an individual introductory meeting with staff including psychiatric and somatic examination, self-assessment scales for symptoms and quality of life, and blood samples. The training period ends with a meeting with staff with follow-up on the parameters.

SUMMARY:
"Braining" is a clinical method for physical exercise as adjunctive therapy in psychiatric care. The core components are personnel-led group training sessions and motivating contact with psychiatric staff, as well as measurement and evaluation before and after the training period of 12 weeks.

Objective. This study aims to describe the clinical and demographic variables in the population of patients who participated in Braining 2017-2020, investigate the feasibility of Braining, and analyse perceived short-term effects and side effects of Braining regarding psychiatric and somatic symptoms.

Method. The project is a retrospective, descriptive study. Patients at Psykiatri Sydväst (PSV, Psychiatric Clinic Psychiatry Southwest, Stockholm) who participated in Braining 2017-2020 during at least 3 training sessions, will be asked for inclusion. Medical and demographic data, as well as patient treatment evaluations, are already available in medical records.

Additionally, an extended 2-year long-term follow-up will be carried out. This includes blood and hair sample, physical examination as well as qualitative interviews with a representative subgroup.

DETAILED DESCRIPTION:
The method "Braining" is a clinical invention that helps patients to initiate and execute physical exercise (PE) regularly in psychiatric care. The core components are basic high performance group training sessions and motivational work led by the psychiatric staff. Braining is used as add-on treatment to regular psychiatric care (treatment as usual; TAU) and is included in the patient care plan. Braining is unique in that it:

1. Includes trained psychiatric clinical staff leading group exercise sessions together with patients from both out- and inpatient ward units in daily, high endurance group training sessions.
2. Is included in regular healthcare fee (free of charge).
3. Includes a motivational and educational visit (as either a group seminar or as an individual visit) at the start and end of a training period; usually 12 weeks.
4. Includes regular measurements (self-assessment questionnaires, blood samples, physical and mental health examination and education before and after the twelve week training period).
5. Includes short individual motivating visits before every training session, including assessment of day shape and fitness to participate.

The scientific purpose of the project is to:

* Describe clinical and demographic variables in patients participating in Braining 2017-2020.
* Investigate the feasibility of the Braining method (PE together with staff as adjunctive therapy in Psychiatric care).
* Analyse perceived short-term effects and side effects of Braining regarding psychiatric and somatic symptoms (degree of psychiatric symptoms, changes in molecular and cardiovascular parameters, lifestyle patterns, level of functioning and perceived quality of life). Also, if possible, provide an estimate of what long-term effects that might be expected in coming long-term clinical follow-ups.
* Investigate patients' long term experience of Braining participation through qualitative interviews as well as analyse status and change of biomolecular markers two years after inclusion.

Specific goals:

All patients at PSV who participated in Braining 2017-2020 during at least 3 training sessions and do not meet the exclusion criteria will be asked for inclusion. For this population the investigators plan to describe:

* Demographic and medical variables (such as diagnosis, age, gender, functional level, staff-assessed severity of psychiatric disease, self-assessment scales for symptoms of depression, mania / hypomania, and anxiety, self-assessed health-related quality of life, degree of sick leave, ongoing pharmacological treatment, ongoing CBT (cognitive behavioral therapy), need for emergency visits, inpatient care, suicidal attempts).
* Feasibility of the Braining method. Evaluation of the degree of participation in Braining (such as number of training sessions performed, participation over time, differences between subgroups, possible incidents) as well as the participants' experience of Braining (based on surveys and follow-up interviews: positive or negative subjective assessments of the method, to what extent is the method recommended to other patients). Adverse events.
* Differences before and after Braining in terms of statistically significant change in [I] degree of psychiatric symptoms and function, [II] cardio metabolic factors such as blood pressure, BMI, waist measurement, weight, [III] molecular parameters such as serum concentration of blood lipids, fasting blood sugar, HbA1c, CRP, [IV] health-related quality of life, [V] level of social function (such as work/study/sick leave) and care needs (such as need of inpatient care, medicine, emergency visits), [VI] assessed severity of psychiatric disorder, [VII] lifestyle patterns such as exercise, sleep, diet, substance use.

ELIGIBILITY:
Inclusion Criteria:

• ≥3 training sessions during the years 2017-2020

Exclusion Criteria:

* <3 training sessions during the years 2017-2020
* Does not speak Swedish
* Care in accordance with the Compulsory Mental Care Act (Lagen om psykiatrisk tvångsvård, LPT)
* Total lack of data at the start of participation in Braining
* Deceased

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Braining 2017-2020 was primarily open for patients with a main or secondary diagnosis in affective illness or anxiety syndromes, or with depression, anxiety, sleep disturbance or stress as sub-symptoms of other psychiatric disorder.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-12-20 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Descriptives of the population | 2017-2020
  The investigators plan to describe the population from a socioeconomic, demographic and medical perspective. The study design is observational, and therefore not hypothesis-driven. The study design is is not a clinical trial.
Feasibility - The population´s participation in Braining | 2017-2020
  The population's participation in terms of number of training sessions, participation over time, differences between subgroups. General description of how the participants experienced the method (common positive or negative subjective assessments of the method, the extent to which the method is recommended to other patients), based on the participants' treatment evaluations. Adverse events. The study design is observational, and therefore not hypothesis-driven. The study design is not a clinical trial.
PHQ-9 (Patient Health Questionnaire - 9 items) | At the individual's start of participation in Braining (T0)
  Self-assessment of symptoms of depression. Symptom assessment tool that measures health using nine items on 4-point scales and a 4-point scale for impact on daily life. Score 0-27. A higher value indicates worse symptoms of depression.
PHQ-9 (Patient Health Questionnaire - 9 items) | At inclusion (Ti)
  Self-assessment of symptoms of depression. Symptom assessment tool that measures health using nine items on 4-point scales and a 4-point scale for impact on daily life. Score 0-27. A higher value indicates worse symptoms of depression.
GAD-7 (Generalised Anxiety Disorder Assessment - 7 items) | At the individual's start of participation in Braining (T0)
  Self-assessment of symptoms of generalised anxiety. Symptom assessment tool that measures seven anxiety symptoms on 4-point scales. Score 0-21. A higher value indicates worse symptoms of general anxiety.
GAD-7 (Generalised Anxiety Disorder Assessment - 7 items) | At inclusion (Ti)
  Self-assessment of symptoms of generalised anxiety. Symptom assessment tool that measures seven anxiety symptoms on 4-point scales. Score 0-21. A higher value indicates worse symptoms of general anxiety.
CGI-S (Clinical Global Impressions - Severity Scale) | At the individual's start of participation in Braining (T0)
  A one-item clinician assessed measure which evaluates the severity of psychopathology from 1 to 7, where 1 is 'normal' and 7 is 'among the most extremely ill patients' by the question "Considering your total clinical experience with this particular population, how mentally ill is the patient at this time?".
CGI-S (Clinical Global Impressions - Severity Scale) | At inclusion (Ti)
  A one-item clinician assessed measure which evaluates the severity of psychopathology from 1 to 7, where 1 is 'normal' and 7 is 'among the most extremely ill patients' by the question "Considering your total clinical experience with this particular population, how mentally ill is the patient at this time?".
Blood pressure | At the individual's start of participation in Braining (T0)
  Blood pressure, systolic and diastolic, mmHg
Blood pressure | At inclusion (Ti)
  Blood pressure, systolic and diastolic, mmHg
BMI (Body Mass Index) | At the individual's start of participation in Braining (T0)
  Weight in kg divided by the square of height in m
BMI (Body Mass Index) | At inclusion (Ti)
  Weight in kg divided by the square of height in m
FBS (Fasting Blood Sugar) | At the individual's start of participation in Braining (T0)
  Fasting blood sugar, mmol/L
FBS (Fasting Blood Sugar) | At inclusion (Ti)
  Fasting blood sugar, mmol/L
EQ-5D ( EQ-5D™ is a trade mark of the EuroQol Group) | At the individual's start of participation in Braining (T0)
  Self-assessment instrument for describing and valuing health. Defines health in terms of five dimensions: Mobility, Self-Care, Usual Activities, Pain/Discomfort, and Anxiety/Depression. Also included is an overall health rating on a 0-100 hash-marked, vertical visual analogue scale (EQ-VAS). Assessment the scores from the descriptive component can be reported as a five digit number ranging from 11111 (full health) to 33333 (worst health). A number of methods exist for analysing these five digit profiles. However, frequently they are converted to a single utility index using country specific value sets. A higher index number indicates a poorer self-assessed health.
EQ-5D ( EQ-5D™ is a trade mark of the EuroQol Group) | At inclusion (Ti)
  Self-assessment instrument for describing and valuing health. Defines health in terms of five dimensions: Mobility, Self-Care, Usual Activities, Pain/Discomfort, and Anxiety/Depression. Also included is an overall health rating on a 0-100 hash-marked, vertical visual analogue scale (EQ-VAS). Assessment the scores from the descriptive component can be reported as a five digit number ranging from 11111 (full health) to 33333 (worst health). A number of methods exist for analysing these five digit profiles. However, frequently they are converted to a single utility index using country specific value sets. A higher index number indicates a poorer self-assessed health.

SECONDARY OUTCOMES:
AS-18 (Affective Self Assessment Scale - 18 items) | At the individual's start of participation in Braining (T0)
  Self-assessment of symptoms of depression and hypomania/mania. 9 items for depression and 9 items for mania. Score 0-72. A score of over 10 on the depressive or manic/hypomanic subscale should give rise to suspicion of ongoing depression and hypomania/mania respectively. Scores of over 10 on both the depressive and manic/hypomanic scale at the same time give may indicate an affective mixed state.
AS-18 (Affective Self Assessment Scale - 18 items) | At inclusion (Ti)
  Self-assessment of symptoms of depression and hypomania/mania. 9 items for depression and 9 items for mania. Score 0-72. A score of over 10 on the depressive or manic/hypomanic subscale should give rise to suspicion of ongoing depression and hypomania/mania respectively. Scores of over 10 on both the depressive and manic/hypomanic scale at the same time give may indicate an affective mixed state.
YMRS (Young Ziegler Mania Rating Scale) | At the individual's start of participation in Braining (T0)
  Interviewer-rated scale. Includes 11 items; seven are rated from 0 (absent) to 4; four from 0 to 8; total scores range from 0 to 60. A higher value indicates worse symptoms of hypomania/mania.
YMRS (Young Ziegler Mania Rating Scale) | At inclusion (Ti)
  Interviewer-rated scale. Includes 11 items; seven are rated from 0 (absent) to 4; four from 0 to 8; total scores range from 0 to 60. A higher value indicates worse symptoms of hypomania/mania.
LSAS (Liebowitz Social Anxiety Scale) | At the individual's start of participation in Braining (T0)
  Self-assessment of symptoms of social anxiety. Comprises 24 social situations that are each rated for level of fear and avoidance. Score (including both subscales) 0-144. A higher value indicates worse symptoms of social anxiety.
LSAS (Liebowitz Social Anxiety Scale) | At inclusion (Ti)
  Self-assessment of symptoms of social anxiety. Comprises 24 social situations that are each rated for level of fear and avoidance. Score (including both subscales) 0-144. A higher value indicates worse symptoms of social anxiety.
PDSS (Panic Disorder Severity Scale) | At the individual's start of participation in Braining (T0)
  Self-assessment of symptoms of panic disorder. The 7-item scale assesses the frequency of panic attacks, distress during panic attacks, anticipatory anxiety, agoraphobic fear and avoidance, body-sensation fear and avoidance, and impairment in work and social functioning on 5-point scales (0-4). Score 0-28. A higher value indicates worse symptoms of panic disorder.
PDSS (Panic Disorder Severity Scale) | At inclusion (Ti)
  Self-assessment of symptoms of panic disorder. The 7-item scale assesses the frequency of panic attacks, distress during panic attacks, anticipatory anxiety, agoraphobic fear and avoidance, body-sensation fear and avoidance, and impairment in work and social functioning on 5-point scales (0-4). Score 0-28. A higher value indicates worse symptoms of panic disorder.
AUDIT (Alcohol Use Disorders Identification Test) | At the individual's start of participation in Braining (T0)
  Self-report instrument used to identify problematic use of alcohol. Value 0-40. A score of 8 for men and 6 for women is usually set as the clinical cut-off for problematic use. A higher value indicates more problematic use.
AUDIT (Alcohol Use Disorders Identification Test) | At inclusion (Ti)
  Self-report instrument used to identify problematic use of alcohol. Value 0-40. A score of 8 for men and 6 for women is usually set as the clinical cut-off for problematic use. A higher value indicates more problematic use.
DUDIT (Drug Use Disorders Identification Test) | At the individual's start of participation in Braining (T0)
  Self-report instrument used to identify problems with illegal drugs and/or prescription drugs. Value 0-44. A score of 6 for men and 2 for women is usually set as the clinical cut-off for harmful use. A higher value indicates more problematic use.
DUDIT (Drug Use Disorders Identification Test) | At inclusion (Ti)
  Self-report instrument used to identify problems with illegal drugs and/or prescription drugs. Value 0-44. A score of 6 for men and 2 for women is usually set as the clinical cut-off for harmful use. A higher value indicates more problematic use.
HR (Heart Rate) | At the individual's start of participation in Braining (T0)
  Heart rate, bpm
HR (Heart Rate) | At inclusion (Ti)
  Heart rate, bpm
Waist circumference | At the individual's start of participation in Braining (T0)
  Waist circumference, cm
Waist circumference | At inclusion (Ti)
  Waist circumference, cm
Blood lipids | At the individual's start of participation in Braining (T0)
  Total cholesterol, LDL cholesterol, HDL cholesterol, triglycerides, mmol/L
Blood lipids | At inclusion (Ti)
  Total cholesterol, LDL cholesterol, HDL cholesterol, triglycerides, mmol/L
HbA1c | At the individual's start of participation in Braining (T0)
  Hemoglobin A1c, glycated hemoglobin, mmol/mol
HbA1c | At inclusion (Ti)
  Hemoglobin A1c, glycated hemoglobin, mmol/mol
CRP | At the individual's start of participation in Braining (T0)
  C-reactive protein, measurement of inflammation and infection, mmol/L
CRP | At inclusion (Ti)
  C-reactive protein, measurement of inflammation and infection, mmol/L
WHODAS 2.0 (WHO Disability Assessment Schedule) | At the individual's start of participation in Braining (T0)
  Self-assessment of disability. Covering six domains concerning functioning: cognitive, mobility, self-care, getting along with people, life activities, and social participation. The summary score is converted into a metric ranging from 0 to 100 (where 0 = no disability; 100 = full disability).
WHODAS 2.0 (WHO Disability Assessment Schedule) | At inclusion (Ti)
  Self-assessment of disability. Covering six domains concerning functioning: cognitive, mobility, self-care, getting along with people, life activities, and social participation. The summary score is converted into a metric ranging from 0 to 100 (where 0 = no disability; 100 = full disability).
Occupational status | At the individual's start of participation in Braining (T0)
  Employment, unemployment, sick leave, early retirement, retirement pension
Occupational status | At inclusion (Ti)
  Employment, unemployment, sick leave, early retirement, retirement pension
Acceptability of treatment method among patients | Follow-up 2 years after inclusion
  Semi-structured interviews. Qualitative technique that explores patients' experiences. No scale.

CONTACTS AND LOCATIONS:
Overall Officials: Lina Martinsson, MD, PhD, Principal Investigator — Karolinska Institute and Region Stockholm
Locations (1):
- Region Stockholm, Psykiatri Sydväst (Psychiatric Clinic Psychiatry Southwest), Stockholm, Stockholm County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Whiteford HA, Degenhardt L, Rehm J, Baxter AJ, Ferrari AJ, Erskine HE, Charlson FJ, Norman RE, Flaxman AD, Johns N, Burstein R, Murray CJ, Vos T. Global burden of disease attributable to mental and substance use disorders: findings from the Global Burden of Disease Study 2010. Lancet. 2013 Nov 9;382(9904):1575-86. doi: 10.1016/S0140-6736(13)61611-6. Epub 2013 Aug 29. PMID 23993280
- [Background] Goodwin GM, Haddad PM, Ferrier IN, Aronson JK, Barnes T, Cipriani A, Coghill DR, Fazel S, Geddes JR, Grunze H, Holmes EA, Howes O, Hudson S, Hunt N, Jones I, Macmillan IC, McAllister-Williams H, Miklowitz DR, Morriss R, Munafo M, Paton C, Saharkian BJ, Saunders K, Sinclair J, Taylor D, Vieta E, Young AH. Evidence-based guidelines for treating bipolar disorder: Revised third edition recommendations from the British Association for Psychopharmacology. J Psychopharmacol. 2016 Jun;30(6):495-553. doi: 10.1177/0269881116636545. Epub 2016 Mar 15. PMID 26979387
- [Background] Aylett E, Small N, Bower P. Exercise in the treatment of clinical anxiety in general practice - a systematic review and meta-analysis. BMC Health Serv Res. 2018 Jul 16;18(1):559. doi: 10.1186/s12913-018-3313-5. PMID 30012142
- [Background] Melo MC, Daher Ede F, Albuquerque SG, de Bruin VM. Exercise in bipolar patients: A systematic review. J Affect Disord. 2016 Jul 1;198:32-8. doi: 10.1016/j.jad.2016.03.004. Epub 2016 Mar 15. PMID 26998794
- [Background] Strohle A, Graetz B, Scheel M, Wittmann A, Feller C, Heinz A, Dimeo F. The acute antipanic and anxiolytic activity of aerobic exercise in patients with panic disorder and healthy control subjects. J Psychiatr Res. 2009 Aug;43(12):1013-7. doi: 10.1016/j.jpsychires.2009.02.004. Epub 2009 Mar 16. PMID 19289240
- [Background] Hofmann SG, Asnaani A, Vonk IJ, Sawyer AT, Fang A. The Efficacy of Cognitive Behavioral Therapy: A Review of Meta-analyses. Cognit Ther Res. 2012 Oct 1;36(5):427-440. doi: 10.1007/s10608-012-9476-1. Epub 2012 Jul 31. PMID 23459093
- [Background] Shafran R, Clark DM, Fairburn CG, Arntz A, Barlow DH, Ehlers A, Freeston M, Garety PA, Hollon SD, Ost LG, Salkovskis PM, Williams JM, Wilson GT. Mind the gap: Improving the dissemination of CBT. Behav Res Ther. 2009 Nov;47(11):902-9. doi: 10.1016/j.brat.2009.07.003. Epub 2009 Aug 6. PMID 19664756
- [Background] Layard R, Clark DM. Why More Psychological Therapy Would Cost Nothing. Front Psychol. 2015 Nov 25;6:1713. doi: 10.3389/fpsyg.2015.01713. eCollection 2015. No abstract available. PMID 26635648
- [Background] Wolitzky-Taylor K, Zimmermann M, Arch JJ, De Guzman E, Lagomasino I. Has evidence-based psychosocial treatment for anxiety disorders permeated usual care in community mental health settings? Behav Res Ther. 2015 Sep;72:9-17. doi: 10.1016/j.brat.2015.06.010. Epub 2015 Jul 2. PMID 26159908
- [Background] Abosi O, Lopes S, Schmitz S, Fiedorowicz JG. Cardiometabolic effects of psychotropic medications. Horm Mol Biol Clin Investig. 2018 Jan 10;36(1):/j/hmbci.2018.36.issue-1/hmbci-2017-0065/hmbci-2017-0065.xml. doi: 10.1515/hmbci-2017-0065. PMID 29320364
- [Background] Ekelund U, Tarp J, Steene-Johannessen J, Hansen BH, Jefferis B, Fagerland MW, Whincup P, Diaz KM, Hooker SP, Chernofsky A, Larson MG, Spartano N, Vasan RS, Dohrn IM, Hagstromer M, Edwardson C, Yates T, Shiroma E, Anderssen SA, Lee IM. Dose-response associations between accelerometry measured physical activity and sedentary time and all cause mortality: systematic review and harmonised meta-analysis. BMJ. 2019 Aug 21;366:l4570. doi: 10.1136/bmj.l4570. PMID 31434697
- [Background] Cooney GM, Dwan K, Greig CA, Lawlor DA, Rimer J, Waugh FR, McMurdo M, Mead GE. Exercise for depression. Cochrane Database Syst Rev. 2013 Sep 12;2013(9):CD004366. doi: 10.1002/14651858.CD004366.pub6. PMID 24026850
- [Background] Helgadottir B, Forsell Y, Ekblom O. Physical activity patterns of people affected by depressive and anxiety disorders as measured by accelerometers: a cross-sectional study. PLoS One. 2015 Jan 13;10(1):e0115894. doi: 10.1371/journal.pone.0115894. eCollection 2015. PMID 25585123
- [Background] Mead GE, Morley W, Campbell P, Greig CA, McMurdo M, Lawlor DA. Exercise for depression. Cochrane Database Syst Rev. 2008 Oct 8;(4):CD004366. doi: 10.1002/14651858.CD004366.pub3. PMID 18843656
- [Background] Rimer J, Dwan K, Lawlor DA, Greig CA, McMurdo M, Morley W, Mead GE. Exercise for depression. Cochrane Database Syst Rev. 2012 Jul 11;(7):CD004366. doi: 10.1002/14651858.CD004366.pub5. PMID 22786489
- See also: Swedish Professional Associations for Physical Activity (Yrkesföreningar för Fysisk Aktivitet, YFA). 2021. Physical Activity in the Prevention and Treatment of Disease (FYSS). 2021. — http://www.fyss.se
- See also: World Health Organization. (2020). WHO guidelines on physical activity and sedentary behaviour: at a glance. World Health Organization. — https://apps.who.int/iris/handle/10665/337001
- See also: 2018 Physical Activity Guidelines Advisory Committee. 2018 Physical Activity Guidelines Advisory Committee Scientific Report. Washington, DC: U.S. Department of Health and Human Services, 2018 — https://health.gov/sites/default/files/2019-09/PAG_Advisory_Committee_Report.pdf